CLINICAL TRIAL: NCT03881969
Title: Does Paying Subjects to Participate in Research Improve Recruitment and Increase the Proportion of Socially Deprived and Elderly Participants?
Brief Title: Does Paying Subjects to Participate in Research Improve Recruitment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012 CV01
Record Dates: First submitted 2016-01-07; First posted 2019-03-20 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Diseases
Keywords: Trial Recruitment; Incentive Payment; Patient Demographics
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financial incentive offered (Experimental): Patient offered £100 incentive payment in initial trial invitation letter.
  Interventions: Behavioral: Financial Payment of £100
- No incentive. Payment not offered (Experimental): Patient sent standard trial invitation letter with no offer of incentive payment.
  Interventions: Behavioral: Financial Payment of £100

INTERVENTIONS:
Behavioral: Financial Payment of £100 — No financial payment
  Other Names: No Financial Payment

SUMMARY:
Patient recruitment into clinical trials is a major challenge and the elderly, socially deprived and those with multiple co-morbidities are often under-represented. The idea of paying patients an incentive to participate in research is controversial and evidence is needed to evaluate this as a recruitment strategy. This study aims to assess the impact on recruitment into five current clinical trials of a £100 incentive payment and whether this payment will attract more elderly and socially deprived patients.

DETAILED DESCRIPTION:
In the UK, it is already common practice to reimburse out-of-pocket expenses eg travelling expenses and parking charges to patients participating in clinical research studies, but not to give any other incentives. This contrasts with healthy volunteer studies where financial payments are often made to encourage participation in studies.

There are few data on how payments to patients in the UK would influence the recruitment and demographic structure of patients recruited to clinical research studies.

The single biggest cost of clinical trials in the UK is the cost of recruiting suitable subjects. The Academy of Medical Sciences report on the UK clinical trials environment, "A new pathway for the regulation and governance of health research", provided a comprehensive review of the barriers faced in running clinical trials . However, other barriers to recruitment exist after these hurdles have been overcome. Importantly, in our experience, of 100 suitable subjects identified as suitable to be entered into a study only about 14% are actually randomised. Most of the identified suitable subjects do not reply to invitation letters from their doctor and some patients who do reply decline the invitation to participate. Campaigns to engage the public on the importance of research have had modest effects on improving the awareness about trials but no measurable effect on willingness to participate .

An important finding is that those subjects who do participate in clinical trials usually have much lower rates of events than predicted from observational data. This is probably because trials attract subjects who care about their own health and the health of others and these subjects exhibit good 'health behaviour'. Those subjects with less good health behaviour and who constitute the subjects who suffer more consequences from their disorders in the real world, do not participate in trials as readily. The result is that trial participants tend to be middle class, middle aged, low risk subjects. These subjects are unrepresentative of the population at large or the population who will eventually get most of the prescribing (lower class, elderly and high risk). In addition, including only low risk subjects may result in studies being abandoned because the low event rates make achieving a statistically reliable result futile.

How can we address this issue within an ethical framework?

The findings from one trial currently running casts some light on this issue. The Streamlined Celecoxib versus standard therapy Outcome Trial (SCOT) is currently running in both the UK and Denmark. Trial recruitment in Denmark is significantly better than in the Scotland. We think that this is because in Denmark, all patients pay the full price for their medications and trial participation means that they get their medication free. In Scotland where recruitment is lower, all prescriptions are free anyway so there is no such incentive. Thus there appears to be a financial incentive for Danish patients to participate.

The present proposal seeks to study the effect of payments on recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for inclusion in one of the 5 clinical trials involved in the paying patients trial.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Patient response to initial invitation letter | On Study completion Approx 1 year
  Number of positive responses to the initial invitation to participate in a clinical trial letter as determined by whether or not the patient was offered £100 incentive payment.

SECONDARY OUTCOMES:
Recruitement of elderly and socially deprived patients | Through study completion Approx 1 year
  To determine whether the offer of £100 incentive would result in increased recruitment of elderly or socially deprived patients. Social deprivation determined by postcode and Scottish Index of Multiple Deprivation (SIMD) score.

IPD SHARING:
Plan to Share IPD: No